CLINICAL TRIAL: NCT03812913
Title: Neuropsychological Assessment of Children and Adolescents With Turner Syndrome
Acronym: ENEAST
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2018-A01478-47
Record Dates: First submitted 2018-10-29; First posted 2019-01-23 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Turner Syndrome; Isolated Growth Hormone Deficiency; Cognitive Functions; Social Cognition; Pediatrics
Keywords: Turner syndrome; Cognitive Functions; Social Cognition; Pediatrics
MeSH Terms: conditions — Turner Syndrome; Dwarfism, Pituitary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Turner Syndrome: * 35 girls with Turner syndrome (except patients with part of a Y chromosome in their karyotype and r(X) cases).
  * age : 7 years -16 years and 11 months.
  * Psychological evaluation of cognition, social cognition and affective cognition
  Interventions: Behavioral: psychological evaluation
- isolated GHD: * 35 girls with isolated Growth Hormone Deficiency (GHD).
  * age : 7 years -16 years and 11 months.
  * Psychological evaluation of cognition, social cognition and affective cognition
  Interventions: Behavioral: psychological evaluation

INTERVENTIONS:
Behavioral: psychological evaluation — * Neuropsychological and experimental tasks will assess cognitive and socio-cognitive functions.
  * Questionnaires will assess psychoaffective aspects (depression, anxiety, self-esteem), and social and behavioral functioning.

SUMMARY:
Turner syndrome (TS) is a rare chromosomal disorder characterized by partial or complete loss of one of the X chromosomes that affects about one in every 2000 female babies born. These young patients described difficulties making friends, understanding others' emotions and intentions, and controlling their own emotions. Difficulties in these domains could led to social withdrawal, to reduced social skills and could have a significant impact on self esteem and mental health as well as on long-term academic and social functioning in affected individuals. The purpose of this project is to identify functional and dysfunctional cognitive and socio-cognitive abilities in these young patients which could account social difficulties described by some of them and their family. To this end, 35 girls with TS and 35 girls with isolated growth hormone deficiency and normal cerebral MRI will be recruited. Subjects will be 7 to 16 years and 11 months of age. Socio-cognitive and cognitive functions will be assessed with neuropsychological and experimental tasks. Questionnaires completed by patient, parents or teacher, will evaluate social and behavioral functioning.

DETAILED DESCRIPTION:
Cross-sectional study (2 groups : Turner syndrome, isolated growth hormone deficiency), not randomized, controlled, associating several specialized centers in endocrine diseases.

The pediatric endocrinologist of the participating centers will contact parents of each patient or voluntary child/adolescent in order to inform them of the study.

The visit of inclusion will take place in the participant center during a routine monitoring visit.

The first visit (V1) will take place immediately after the visit of inclusion in order to avoid a specific displacement for the needs for the study. The second visit (V2) will take place in participant's home. Each visit (V1 and V2) will last half-day. The period between V1 and V2 will be three months maximum.

The visits V1 and V2 will be carried out by neuropsychologists of the Laboratoire de Psychologie des Pays de la Loire (LPPL - EA 4638).

ELIGIBILITY:
INCLUSION CRITERIA

Turner syndrome group :

* girls with diagnosed Turner syndrome.

Isolated GHD group :

* girls with diagnosed isolated growth hormone deficiency

All participants :

* age between 7 years to 16 years and 11 months.
* informed consent signed by the participant and her parents (or her legal representatives)
* being registered in the national social security system

EXCLUSION CRITERIA :

Turner syndrome group :

* patients with chronic pathology other than Turner syndrome.
* karyotype : part of a Y chromosome and r(X) cases.
* medical treatment other than those usually prescribed in patients with Turner syndrome.

Isolated GHD group :

* patients with chronic pathology other than isolated growth hormone deficiency.
* medical treatment other than those usually prescribed in patients with isolated growth hormone deficiency.

All participants :

* diagnosed intellectual disability (IQ<70) or intellectual giftedness
* history of acquired brain injury
* sensory disturbances (auditory or visual) incompatible with the achievement of neuropsychological tasks.
* insufficient French language proficiency

Ages: 7 Years to 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Study Population: * 35 patients with Turner syndrome
  * 35 patients with isolated growth hormone deficiency
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-09-05 (Actual); Primary Completion 2025-12-05 (Estimated); Study Completion 2025-12-05 (Estimated)

PRIMARY OUTCOMES:
Wechsler Intelligence Scale for Children (WISC-V) | 3 months
  intelligence scale.
Cognitive theory of mind first order | 3 months
  First order theory of mind tasks (Baron-Cohen et al., 1985)
Cognitive theory of mind second order | 3 months
  second-order theory of mind tasks Perner & Wimmer, 1983)
Cognitive theory of mind advanced | 3 months
  advanced theory of mind tasks (Happé, 1994)
Cognitive theory of mind : humor | 3 months
  Humor understanding task
Affective theory of mind : faux pas | 3 months
  Faux pas recognition test (Baron Cohen et al., 1999)
Affective theory of mind : first order | 3 months
  First-order affective theory of mind tasks
Affective theory of mind : second order | 3 months
  Second-order affective theory of mind tasks
Affective theory of mind : emotional inference | 3 months
  Emotional inference for context test
Emotional valence recognition : valence | 3 months
  Emotional valence rating from visual scenes
Facial emotion recogniton | 3 months
  Facial emotion recognition task
Vocal emotion recognition | 3 months
  Emotional prosody recognition task
Emotional regulation | 3 months
  Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA)
Alexithymia | 3 months
  Questionnaire d'alexithymie chez l'enfant (QAE)
Empathy | 3 months
  Interpersonal Reactivity Index (IRI)
Oral Language comprehension abilities 1 | 3 months
  Comprehension of Instructions (NEPSY-II, Korkman et al., 2012)
Oral Language comprehension abilities 2 | 3 months
  Verbal comprehension index (from WISC-V)
Visual and visual-spatial abilities:1 | 3 months
  Arrows subtest (NEPSY-II - Korkman et al., 2012),
Visual and visual-spatial abilities:2 | 3 months
  Picture Puzzles subtest (NEPSY-II - Korkman et al., 2012)
Visual and visual-spatial abilities:3 | 3 months
  Benton Facial Recognition Test (Benton et al., 1983)
Executive abilities-Verbal Working memory 1 | 3 months
  Verbal information updating task
Executive abilities-Visuo-Spatial Working memory 2 | 3 months
  Visuo-spatial information updating task
Executive abilities-Inhibition 1 | 3 months
  Stroop test.
Executive abilities-Inhibition 2 | 3 months
  Tapping test
Executive abilities-Inhibition 3 | 3 months
  non-verbal cancellation task
Executive abilities-Cognitive Flexibility 1 | 3 months
  Verbal fluency task (NEPSY-II Korkman et al., 2012)
Executive abilities-Cognitive Flexibility 2 | 3 months
  Modified Wisconsin Card Sorting Test for children
Executive abilities-Cognitive Flexibility 3 | 3 months
  Trail Making Test
Executive abilities-Higher-order executive functions 1 | 3 months
  script generation task
Executive abilities-Higher-order executive functions 2 | 3 months
  Rey Complex Figure Test : Copy
Executive abilities in daily life | 3 months
  Behavioral Rating Inventory of Executive Functions
Self Esteem | 3 months
  Rosenberg self-esteem scale (1965).
Depression inventory | 3 months
  Depression: Children's Depression Inventory (Kovacks & Beck, 1977).
Anxiety inventory | 3 months
  Revised Children's Manifest Anxiety Scale (Reynolds & Richmond, 1999).
Social desirability | 3 months
  Children's Social Desirability Scale (Crandall et al., 1965)
social adjustment 1 | 3 months
  Conners' Parent Rating Scale-Revised: Short Form (Conners, 1997)
social adjustment 2 | 3 months
  Conners' Teacher Rating Scale-Revised: Short Form (Conners, 1997)
behavioral adjustment | 3 months
  Child Behavior Checklist (Achenbach, 1991).

CONTACTS AND LOCATIONS:
Overall Officials: Régis Coutant, MD PhD, Principal Investigator — UH Angers
Locations (3):
- France (3):
  - CHU Rennes, Rennes, Ile Et Vilaine
  - CHU Nantes, Nantes, Loire Atlantique
  - CHU Angers, Angers, Maine Et Loire

REFERENCES:
- [Background] LoBue V, Thrasher C. The Child Affective Facial Expression (CAFE) set: validity and reliability from untrained adults. Front Psychol. 2015 Jan 6;5:1532. doi: 10.3389/fpsyg.2014.01532. eCollection 2014. PMID 25610415
- [Background] Olszanowski M, Pochwatko G, Kuklinski K, Scibor-Rylski M, Lewinski P, Ohme RK. Warsaw set of emotional facial expression pictures: a validation study of facial display photographs. Front Psychol. 2015 Jan 5;5:1516. doi: 10.3389/fpsyg.2014.01516. eCollection 2014. PMID 25601846
- [Background] Happe FG. An advanced test of theory of mind: understanding of story characters' thoughts and feelings by able autistic, mentally handicapped, and normal children and adults. J Autism Dev Disord. 1994 Apr;24(2):129-54. doi: 10.1007/BF02172093. PMID 8040158
- [Background] Baron-Cohen S, Leslie AM, Frith U. Does the autistic child have a "theory of mind"? Cognition. 1985 Oct;21(1):37-46. doi: 10.1016/0010-0277(85)90022-8. No abstract available. PMID 2934210
- [Background] Wimmer H, Perner J. Beliefs about beliefs: representation and constraining function of wrong beliefs in young children's understanding of deception. Cognition. 1983 Jan;13(1):103-28. doi: 10.1016/0010-0277(83)90004-5. No abstract available. PMID 6681741
- [Background] Gullone E, Taffe J. The Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA): a psychometric evaluation. Psychol Assess. 2012 Jun;24(2):409-17. doi: 10.1037/a0025777. Epub 2011 Oct 24. PMID 22023559